CLINICAL TRIAL: NCT06374238
Title: Peer Support for Adolescents and Emerging Adults With Sickle Cell Pain: Promoting Engagement in Cognitive Behavioral Therapy
Brief Title: Peer Support for Adolescents and Emerging Adults With Sickle Cell Pain
Acronym: PRESENCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Charles Jonassaint, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24040171; UG3HL165839 (NIH)
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-09

CONDITIONS: Pain; Sickle Cell Disease
Keywords: Sickle Cell Disease; Pain management; Cognitive Behavioral Therapy; Wellness
MeSH Terms: conditions — Pain; Anemia, Sickle Cell; Agnosia

STUDY DESIGN:
Intervention Model Description: Three-arm, phase III randomized controlled effectiveness trial. Participants will be randomized 3:3:2 into (1) CBT + peer, (2) self-guided CBT, or (3) UC, stratified by site
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBT w/ Health Coach (Experimental): Group will utilize the Presence app to undergo self CBT for EMA, but with addition of peer health coaches.
  Interventions: Behavioral: CBT+ Health coach
- CBT w/o Health coach (self-guided) (Active Comparator): Group will utilize the Presence app to undergo self-guided CBT for EMA, but without peer health coaches.
  Interventions: Behavioral: CBT w/o Health Coach ( self-guided)
- Usual Care with no access to CBT (Active Comparator): Participants in the UC group will have access to CaRISMA app to complete a daily pain and mood e-diary, daily record of opiate use, and weekly assessment of pain via the Painimation tool. All other care will be at the discretion of their treating provider
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: CBT+ Health coach — Participants will complete the pre-enrollment clinical screening measures (PHQ-9M, GAD-7, and PEG-3) and will repeat those assessments, as well as outcome assessments, at 3 months, 6 months, and 12 months. Participants in CBT w/ Health coach group will engage with the CaRISMA app to complete a daily pain and mood e-diary, daily record of opiate use, and weekly assessment of pain via the Painimation tool. In addition participants will have weekly contact with a peer health coach.
  Other Names: CBT+peer
  Arms: CBT w/ Health Coach
Behavioral: CBT w/o Health Coach ( self-guided) — Participants will complete the pre-enrollment clinical screening measures (PHQ-9M, GAD-7, and PEG-3) and will repeat those assessments, as well as outcome assessments, at 3 months, 6 months, and 12 months. Participants CBT w/o Health coach groups will engage with the CaRISMA app to complete a daily pain and mood e-diary, daily record of opiate use, and weekly assessment of pain via the Painimation tool.
  Arms: CBT w/o Health coach (self-guided)
Behavioral: Usual Care — Participants will complete the pre-enrollment clinical screening measures (PHQ-9M, GAD-7, and PEG-3) and will repeat those assessments, as well as outcome assessments, at 3 months, 6 months, and 12 months. Participants in the UC group will be asked to engage with the CaRISMA app to complete a daily pain and mood e-diary, daily record of opiate use, and weekly assessment of pain via the Painimation tool. All other care will be at the discretion of their treating provider
  Arms: Usual Care with no access to CBT

SUMMARY:
The study, known as the Peer suppoRt for adolescents and Emerging adults with Sickle cell pain: promoting ENgagement in Cognitive behavioral thErapy (PRESENCE), aims to determine the effectiveness of digital CBT in reducing pain, opioid use, and healthcare utilization among AYAs with SCD. It also seeks to understand the role of personalized peer support in enhancing engagement and outcomes of digital CBT interventions.

By leveraging existing infrastructure for delivering virtual peer support interventions, tailored digital CBT programs for individuals with SCD, and partnerships with CBOs, the study aims to provide valuable insights into the feasibility and effectiveness of digital CBT as a pain management strategy for this vulnerable population.

DETAILED DESCRIPTION:
The PRESENCE study aims to address the pressing issue of inadequate pain management for adolescents and young adults (AYAs) with sickle cell disease (SCD). Despite pain being the primary clinical symptom of SCD, effective treatment options are limited, leading to repeated hospitalizations and negative impacts on patients' physical and mental well-being. Opioids, the primary treatment for chronic SCD pain, often fail to provide long-term relief and can result in harmful consequences.

Recognizing the need for alternative approaches, the study hopes to investigate the effectiveness of digital cognitive behavioral therapy (CBT), both with and without personalized peer support delivered through community-based organizations (CBOs). CBT is a well-established method for managing pain in the general population, and digital CBT has shown promise in improving outcomes for individuals with chronic conditions.

The study will involve a multisite, randomized controlled trial with 470 AYAs with SCD who have experienced frequent pain over the past three months. Participants will be randomized into one of three groups:

1. Digital CBT with weekly one-on-one peer support (CBT+peer)
2. Digital CBT without peer support (self-guided CBT)
3. Usual care (UC)

The primary hypotheses of the study are:

Hypothesis 1. AYAs receiving any digital CBT (CBT + peer or self-guided CBT) will have greater improvements in primary pain outcomes (PEG-3 pain intensity and pain interference), and larger decreases in secondary pain outcomes (mean daily pain intensity, pain days, average weekly opioid dose, emergency department visits, hospitalizations) and in psychological outcomes (MoSCS internalized stigma, SCSES sickle cell self-efficacy, PHQ-9M depression, GAD-7 anxiety) than AYAs receiving UC at 6 months post initiation of intervention.

Hypothesis 2. AYAs receiving CBT + peer will have greater improvements in the primary and secondary outcomes described above at 6 months, and greater app engagement, than AYAs receiving self-guided CBT.

This study will have the following assessment time points.

* Baseline = pre-randomization baseline measures

  o Rescreen if SCD verification is not provided within 30 days
* At Randomization = Pain and mood diary using Ecological Momentary Assessment (EMA) assessed daily for a total of 14 days with the first entry occuring immediately prior to randomization/intervention start and then continuing daily post-randomization
* 3-month = end of intervention period assessment 90 days (3 months) post -randomization
* 6-month = primary endpoint 180 days (6 months) post-randomization
* 12-month = long-term endpoint 365 days (12 months) post-randomization

The study intervention and EMA data collection is performed via an iOS and Android application called CaRISMA that will be called "the app" or the "CaRISMA app" hereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 16 to 30 years of age at time of enrollment
2. Sickle Cell Disease diagnosis of any genotype based on referral or documentation
3. Reports chronic pain (≥4 days/week for past 3 months or more) OR A) Being prescribed pain medication to be taken (≥4 days/week for past 3 months or more) OR B) Taking pain medication (≥4 days/week for past 3 months or more) OR C) Receiving non-pharmaceutical pain treatment (≥4 days/week for past 3 months or more)
4. Access to an iOS or Android mobile device with internet access

Exclusion Criteria:

1. Unable to speak or read English
2. Prior hematopoietic stem cell transplant for sickle cell disease

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 470 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Determine the effectiveness of any digital CBT (CBT + peer or self-guided CBT) vs usual care (UC) to improve pain intensity for AYAs with SCD and chronic pain | Baseline and 6 months
  Mean change in pain intensity as measured by the Pain, Enjoyment of Life and General Activity (PEG-3) scale. Item 1 asks individuals to rate their pain, on average, over the past week, using a 0-10 rating scale.
Determine the effectiveness of any digital CBT (CBT + peer or self-guided CBT) vs usual care (UC) to improve pain interference for AYAs with SCD and chronic pain | Baseline and 6 months
  Mean change in pain interference as measured by the PEG-3 items 2 and 3 that ask individuals to rate how pain has interfered with their enjoyment and general activities, in the past week, using a 0-10 rating scale.

SECONDARY OUTCOMES:
Determine the effectiveness of CBT+ peer vs. self-guided CBT to improve pain intensity for AYAs with SCD and chronic pain | Baseline and 6 months
  Mean change in pain intensity as measured by the PEG-3
Determine the effectiveness of CBT+ peer vs. self-guided CBT to improve pain interference for AYAs with SCD and chronic pain | Baseline and 6 months
  Mean change in pain interference as measured by the PEG-3
Determine the sustained effectiveness of any digital CBT (CBT + peer or self-guided CBT) vs UC to improve pain intensity for AYAs with SCD and chronic pain | Baseline and 12 months
  Mean change in pain intensity as measured by the PEG-3
Determine the sustained effectiveness of any digital CBT (CBT + peer or self-guided CBT) vs UC to improve pain interference for AYAs with SCD and chronic pain | Baseline and 12 months
  Mean change in pain interference as measured by the PEG-3
Determine the sustained effectiveness of CBT+ peer vs self-guided CBT to improve pain intensity of AYAs with SCD and chronic pain | Baseline and 12 Months
  Mean change in pain intensity as measured by the PEG-3
Determine the sustained effectiveness of CBT+ peer vs self-guided CBT to improve pain interferences of AYAs with SCD and chronic pain | Baseline and 12 Months
  Mean change in pain interference as measured by the PEG-3

CONTACTS AND LOCATIONS:
Overall Officials: Charles Jonassaint, PhD, Principal Investigator — University of Pittsburgh; Ana Radovic, MD, Principal Investigator — University of Pittsburgh; Alicia Colvin, PhD, Principal Investigator — University of Pittsburgh
Locations (14):
- United States (14):
  - University of South Alabama Medical Center, Mobile, Alabama
  - UCLA Mattel Children's Hospital Ronald Reagan Hospital, Los Angeles, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The Regents of the University of Michigan, Ann Arbor, Michigan
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Weil Cornell Medical College, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Wake Forest Baptist Hospital, Durham, North Carolina
  - East Carolina University Health Medical Center, Greenville, North Carolina
  - UPMC University of Pittsburgh Classical Hematology Adult Clinic, Pittsburgh, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No